CLINICAL TRIAL: NCT01886001
Title: Topical Umbilical Cord Care for the Prevention of Colonization and Invasive Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, David A Kaufman, Medical Doctor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16396
Record Dates: First submitted 2013-06-17; First posted 2013-06-25 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Colonization
Keywords: Newborn Intensive Care Unit; Neonatal Intensive Care Unit; Colonization; Line Colonization; Umbilical line; Umbilical Cord Care
MeSH Terms: interventions — Povidone-Iodine; Chlorhexidine; chlorhexidine gluconate; Ethanol; Poloxamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Povidone-Iodine (Betadine) (Experimental): Umbilical stump care. Povidone-Iodine, USP, Swabstick Singles, applied once a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Povidone-Iodine
- Chlorhexidine (Experimental): Umbilical stump care. ChloraPrep® Chlorhexidine Gluconate 2% w/v; 70% Isopropyl Alcohol v/v Swabstick Single, applied once a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Chlorhexidine
- Pluronic (Experimental): Umbilical stump care. Pluronic gel - (F68, Polymyxin, Nystatin, Nitrofurantoin )applied once a day to cord stump while umbilical line(s) are in place
  Interventions: Drug: Pluronic
- Control (no application) (Sham Comparator): Control arm, no product is applied, which is standard of care.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Povidone-Iodine — Umbilical stump care. Povidone-Iodine, USP, Swabstick Singles, applied once a day to cord stump while umbilical line(s) are in place
  Other Names: Betadine
  Arms: Povidone-Iodine (Betadine)
Drug: Chlorhexidine — Umbilical stump care. Chlorhexidine Gluconate 2% w/v; 70% Isopropyl Alcohol v/v Swabstick Single, applied once a day to cord stump while umbilical line(s) are in place
  Other Names: ChloraPrep®; Chlorhexidine Gluconate 2% w/v;70% Isopropyl Alcohol
  Arms: Chlorhexidine
Drug: Pluronic — Umbilical stump care. Pluronic gel - (F68, Polymyxin, Nystatin, Nitrofurantoin)applied once a day to cord stump while umbilical line(s) are in place
  Other Names: Pluronic Gel
  Arms: Pluronic
Other: Control — No product is applied to cord stump while umbilical line(s) are in place. This is the current standard of care at UVA.
  Arms: Control (no application)

SUMMARY:
Umbilical catheters are necessary for many infants admitted to the Newborn Intensive Care Unit (NICU)and utilized when indicated for up to 7 to 14 days. Bacterial colonization can occur at the umbilical stump and potentially lead to serious bloodstream infections (BSIs). This study is a prospective, randomized controlled feasibility trial to evaluate three types of hygiene products on umbilical line stumps, on the effect of line colonization and subsequent infections. Infants admitted to the NICU with an umbilical line(s) will be randomized into one of four study groups, three products against standard of care (no product). The three products that will be evaluated are currently being used in different capacities for skin care in the UVA NICU. The study hypothesizes that daily topical application of 1 or more antiseptic to the top of the umbilical stump will decrease colonization of the umbilical stump while umbilical lines are in place.

DETAILED DESCRIPTION:
Umbilical catheter associated infections are higher (4.4 vs. 3.4 CLABSIs per 1000 line days) than other central lines such as PICCs and surgically placed CVLin the NICU. (www.CDC.gov - NSHN 2010 Report). Routine care of the skin entry site (e.g. central line dressing care) is standard for other central lines, but there is no standard for care of the umbilical stump while umbilical lines are in place.

In a pilot study to evaluate the relationship of umbilical stump colonization with gestational age, the number of days the catheter was in place, and the type of organisms, colonization was detected in 78% of patients. There was a direct correlation with colonization and line days as well as an inverse relationship with lower gestational age.

This pilot data supported the need for the study of interventions to reduce umbilical stump colonization, which may help decrease blood stream infections (BSIs) associated with umbilical lines in the NICU. The proposed study will evaluate feasibility of once daily product application.

ELIGIBILITY:
Inclusion Criteria:

*≤7 days of life

*Umbilical line(s) in place (UAC and/or UVC)

Exclusion Criteria:

*Not meeting inclusion criteria

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Colonization of umbilical stump | while umbilical lines are in place which is an average of 7 days

SECONDARY OUTCOMES:
Late-onset infection | up to 120 days of life, transfer, death or discharge from NICU
  Late-onset infections include BSI, urinary tract infection (UTI), and meningitis. Catheter associated blood stream infections (CLABSI) for this study will be defined as growth in 1 or more blood cultures of any organism including CONS during or within 48-72 hours of having a central line in place, with signs and symptoms of sepsis, and treated for 7 days. Additionally we will compare the CDC definition of CLABSI between groups, and length of stay (LOS).
contact dermatitis | during intervention which is an average of 7 days
  Skin irritation around the umbilical stump

CONTACTS AND LOCATIONS:
Overall Officials: David A Kaufman, MD, Principal Investigator — UVA School of Medicine
Locations (1):
- Univeristy of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
plan to analyze data and publish